CLINICAL TRIAL: NCT07249034
Title: Impact of Epilepsy on the Brainstem Adenosine Pathway and Its Relation With Arousal and Respiratory Reactivity
Acronym: BRAVE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2025-A01888-41
Record Dates: First submitted 2025-09-26; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-09

CONDITIONS: Epilepsy; Drug-resistant Focal Epilepsy; Healthy Controls
Keywords: Epilepsy; adenosine pathway; respiratory reactivity; PET-MRI; [18F]CPFPX
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with drug-resistant epilepsy (Experimental): Diagnosis of refractory focal epilepsy or of refractory idiopathic generalized epilepsy, as defined by the International League Against Epilepsy.
  The following procedures will be carried out as part of the research:
  * Hypercapnic challenge
  * PET/MRI acquisition with [18F]-CPFPX Baseline (0-70 min) Hypercapnic challenge (Breath holding) (70-100 min) Return to equilibrium (100-120 min)
  Interventions: Procedure: 1 Hypercapnic challenge while participant is awake; Procedure: PET/MRI acquisition
- Healthy subjects (Experimental): Selection of healthy subjects will be performed to ensure age and sex matching.
  The following procedures will be carried out as part of the research:
  * Hypercapnic challenge
  * PET/MRI acquisition with [18F]-CPFPX Baseline (0-70 min) Hypercapnic challenge (Breath holding) (70-100 min) Return to equilibrium (100-120 min)
  Interventions: Procedure: 1 Hypercapnic challenge while participant is awake; Procedure: PET/MRI acquisition

INTERVENTIONS:
Procedure: 1 Hypercapnic challenge while participant is awake — The healthy patient/subject breathes through the mouth, using a mouthpiece and a nose clip, through a device fitted with a hermetically sealed bag that measures the various parameters of his/her breathing. At the start of the test, the healthy patient/subject breathes ambient air and his or her breathing is measured. Then, after a few minutes, the healthy patient/subject is connected to the bag, breathing in a closed circuit. This causes a gradual increase in carbon dioxide (CO2) in the inspired air. During this time, breathing parameters will be measured and gas exchanges studied with each breath. The test is stopped when the end-tidal carbon dioxide pressure (PetCO2) reaches 60 mm Hg, or in the event of intolerance
Procedure: PET/MRI acquisition — The PET/MRI acquisition will be organized into 3 parts for a total duration of 120 minutes from the injection of the radiotracer
  1. Baseline (0-70 min)
  2. Respiratory challenge (70-100 min) :
     Subjects will perform three series of expiratory breath holds (six repeats during each run). A green dot will be shown for 30 seconds, indicating that the patient can still breathe normally for 30 seconds. Then, a yellow dot appears for two seconds, indicating that the patient needs to prepare himself for an expiratory BH that shall start at the end of an expiration, and at the end of the two seconds. Then a red dot appears indicating that the patient must hold his breath while being in full expiration or inspiration. The red dot remains until the patient decides to breath again and push a button to alert us of re-breathing. Screen turns black for 60 seconds before another sequence starts (30 sec. green dot).
  3. Return to equilibrium (100-120 min).

SUMMARY:
Despite the continuous development of new antiseizure medications over the past 25 years, 30% of patients with epilepsy suffer from drug-resistant seizures and are at risk of epilepsy-related complications, like cognitive dysfunctions, sleep-disordered breathing or Sudden and Unexpected Death in Epilepsy (SUDEP). SUDEP typically occurs during sleep, after a nocturnal seizure, and primarily results from a postictal central respiratory dysfunction in patients with generalized convulsive seizure (GCS), suggesting that interaction between respiratory dysfunction and sleep state may play a role in its pathophysiology.

Post-mortem data in SUDEP patients showed alteration of neuronal populations involved in respiratory control in the medulla. Accordingly, pharmacologic strategies aimed at reducing the severity of postictal respiratory dysfunction has appeared as one of the most promising way to prevent SUDEP. However, no encouraging result has hitherto been reported.

Interconnections between the complex network that regulates arousal and sleep and the respiratory network are numerous. They primarily include the relation between chemosensitive regulation and arousal system to ensure asphyxia-induced arousal (i.e. arousal to elevated CO2), especially through serotonin (5HT)-dependent connections in brain stem. The link between alterations of the brainstem networks involved in arousal regulation and respiratory dysfunction has not been characterized in patients with epilepsy yet.

Like 5HT, adenosine is deeply implicated in the regulation of sleep and central respiratory control.

Seizures transiently increase adenosine extracellular levels. Adenosine physiological effects in the brain are mediated through the activation of two types of Adenosine receptors (ARs), A1Rs and A2ARs. Extracellular adenosine promotes sleep via A1R-dependant inhibition of glutamatergic neurons in the basal forebrain, but also via A2AR-dependant activation of neurons in the nucleus accumbens. Respiration is also inhibited by A1R and A2AR. Most importantly, it has been shown that drug-resistant epilepsy is associated with long-term alterations of ARs cortical expression. However, whether or not a similar epilepsy-related plasticity of ARs occurs in the brainstem and may participate to chronic arousal and respiratory dysfunction in epilepsy has never been investigated.

Considering the tight interplay between central respiratory control, arousal regulation and brainstem adenosine, the main hypothesis of the BRAVE study is that epilepsy might result in alterations of the distribution of A1Rs in the brainstem structures involved in respiratory regulation and/or arousal control, especially in the brainstem structures involved in respiratory regulation under hypercapnic condition.

The study combines clinical respiratory characterization, morphological, functional and metabolic imaging, using the hybrid simultaneous 3T MRI-PET scanner (Siemens Biograph mMR) of the CERMEP. Combining PET with anatomical and functional MR imaging enables non-invasively in vivo mapping of receptor binding and functional neuronal assessment of a physiological task in the entire brain with high spatial resolution.

Investigators already performed fMRI study of respiratory centers, showing number of functional changes in brainstem regions participating to the central control of respiration, including reduced activation during breath-holding fMRI, in patients with epilepsy. The BRAVE study will use the same respiratory paradigm as the one used in this past study.

PET imaging will be focused on A1R, using [18F]CPFPX, a selective A1R antagonist.

ELIGIBILITY:
Inclusion Criteria:

* For patients

  1. Written informed consent obtained from study subject and ability for study subject to comply with the requirements of the study
  2. Aged 18 to 55 years old
  3. Diagnosis of focal epilepsy or of idiopathic generalized epilepsy, as defined by the International League Against Epilepsy
  4. Diagnosis of refractory epilepsy, as defined by the International League Against Epilepsy
  5. Patients with ≥3 focal to bilateral tonic-clonic seizure (FBTCS) during the past 18 months
  6. For women of childbearing potential, use effective contraception during study participation
* For healthy volunteers

  1. Written informed consent obtained from study subject and ability for study subject to comply with the requirements of the study
  2. Aged 18 to 55 years old
  3. For women of childbearing potential, use effective contraception during study participation

Exclusion Criteria:

* For patients

  1. Ongoing or chronic respiratory and/or cardiac insufficiency
  2. Obstructive sleep-apnea syndrome
  3. Ongoing treatment with selective serotonin reuptake inhibitor
  4. MRI contra-indication (presence of metallic elements, claustrophobia)
  5. Patient treated with vagal nerve stimulation or deep brain stimulation
  6. Pregnant women, women in laboror breastfeeding women, based on declarations at V0
  7. Persons under psychiatric care
  8. Persons deprived of their liberty by a judicial or administrative decision
  9. Adults subject to a legal protection measure (guardianship, curatorship)
  10. Persons not affiliated to a social security scheme or beneficiaries of a similar scheme
  11. Positive urine pregnancy test at V2, if applicable
  12. Hypersensitivity to [18F]-CPFPX
* For healthy volunteers

  1. History of epilepsy
  2. Ongoing or chronic respiratory and/or cardiac insufficiency
  3. Obstructive sleep-apnea syndrome
  4. Ongoing treatment with selective serotonin reuptake inhibitor
  5. MRI contra-indication (presence of metallic elements, claustrophobia)
  6. Pregnant women, women in labor or breastfeeding women, based on declarations at V0
  7. Persons under psychiatric care
  8. Persons deprived of their liberty by a judicial or administrative decision
  9. Adults subject to a legal protection measure (guardianship, curatorship)
  10. Persons not affiliated to a social security scheme or beneficiaries of a similar scheme
  11. Positive urine pregnancy test at V2, if applicable
  12. Hypersensitivity to [18F]-CPFPX

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of the [18F]-CPFPX BPND in the brainstem structures involved in respiratory regulation under hypercapnic condition in patients with drug-resistant epilepsy with the one of healthy subjects | Emission will be acquired over 90 minutes post-injection
  All analyses will be performed on Regions of Interest (ROI), defined as brainstem regions with BOLD activation during BH.
  On the normalized smoothed images, an ANCOVA (analysis of covariance) will be performed, where age, gender and global non-displaceable binding potential (BPND) will be taken into account as covariates of no interest. Statistical parametric maps of the t-statistic (SPM(t)) will be calculated for two contrasts per patient (patient with drug-resistant epilepsy-heathly subjects and heathly subjects-patient with drug-resistant epilepsy) with a threshold of P<0.001 uncorrected at the voxel level; an extent threshold of 100 voxels (of 2mmx2mmx2mm) will be applied at the cluster level

SECONDARY OUTCOMES:
Comparison of the [18F]-CPFPX BPND in the cortical structures involved in respiratory regulation under hypercapnic condition in patients with drug-resistant epilepsy with the one of healthy subjects | Emission will be acquired over 90 minutes post-injection
  All analyses will be performed on Regions of Interest (ROI), defined as cortical regions with BOLD activation during BH.
  On the normalized smoothed images, an ANCOVA (analysis of covariance) will be performed, where age, gender and global non-displaceable binding potential (BPND) will be taken into account as covariates of no interest. Statistical parametric maps of the t-statistic (SPM(t)) will be calculated for two contrasts per patient (patient with drug-resistant epilepsy-heathly subjects and heathly subjects-patient with drug-resistant epilepsy) with a threshold of P<0.001 uncorrected at the voxel level; an extent threshold of 100 voxels (of 2mmx2mmx2mm) will be applied at the cluster level
Evaluating the relation between [18F]-CPFPX BPND in the brainstem structures involved in respiratory regulation under hypercapnic condition and the HCVR slope in patients with drug-resistant epilepsy and in healthy subjects | Emission will be acquired over 90 minutes post-injection
  HCVR measures the increase in minute ventilation (VE) induced by an increase of PETCO2. The HCVR slope, expressed in L/min/mmHg, will be calculated from the linear regression of VE and PETCO2
Comparison of the HCVR slope in patients with drug-resistant epilepsy and in heathly subjects | will be measured during hypercapnic challenges between Day 15 and Day 60 after inclusion
  HCVR measures the increase in minute ventilation (VE) induced by an increase of PETCO2. The HCVR slope, expressed in L/min/mmHg, will be calculated from the linear regression of VE and PETCO2
Evaluating the relation between the HCVR slope and the pattern of BOLD activation during BH in patients with drug-resistant epilepsy and in heathly subjects | will be measured during fMRI acquisition (30 minutes)
  Relation between the HCVR slope and mean % change of the BOLD signal in the regions of Interest (ROI), defined as brainstem or cortical regions with BOLD activation during BH.
Comparing brainstem regional volumes on MRI of patients with drug-resistant epilepsy with the one of healthy subjects | Will ne measured during structural MRI protocol which will include 10 minutes of anatomical imaging
  Gray and white matter volumes will be combined to estimate total brain volume for each subject, which will be used as a covariate in subsequent statistical modelling. Two-sample t tests will used for group comparisons in SPM (patients versus healthy subjects), with age, sex, and total brain volume as covariates. Reported P-values will be family-wise error rate (FWER)-corrected (largest cluster at P < .05). Analysis of relation between VBM and HCVR slope will used Pearson's correlation with age, sex, and total brain volume as covariates. Reported P-values will be family-wise error rate (FWER)-corrected (largest cluster at P < .05).
Evaluating the relation between the brainstem regional volumes on MRI and the HCVR slope in patients with drug-resistant epilepsy and in heathly subjects | Will be measured during structural MRI protocol which will include 10 minutes of anatomical imaging
  Analysis of relation between VBM and HCVR slope will use Pearson's correlation with age, sex, and total brain volume as covariates. Reported P-values will be family-wise error rate (FWER)-corrected (largest cluster at P < .05).
Evaluating the relation between mean daily intake of caffeine (mg/day) and the [18F]-CPFPX BPND in the brainstem and cortical structures | Emission will be acquired over 90 minutes post-injection
  All analyses will be performed on Regions of Interest (ROI), defined as brainstem and cortical regions with BOLD activation during BH.
  Pearson's correlation with age, sex, and global non-displaceable binding potential (BPND) as covariates

CONTACTS AND LOCATIONS:
Overall Officials: Sylvain RHEIMS, PUPH, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon, Bron, France

IPD SHARING:
Plan to Share IPD: No